CLINICAL TRIAL: NCT02990026
Title: Specialty Mental Health Probation in North Carolina
Acronym: SMHP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Department of Public Safety (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-0492; 2015-SM-BX-0004 (Other: UNC)
Record Dates: First submitted 2016-12-06; First posted 2016-12-12 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Mental Illness; Substance Use; Criminal Behavior
MeSH Terms: conditions — Mental Disorders; Substance-Related Disorders; Criminal Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Specialty mental health probation - delivered by probation officers who receive specialized training and ongoing clinical consultation with a licensed mental health professional and who have reduced caseloads of exclusively mentally ill offenders.
  Interventions: Behavioral: Specialty Mental Health Probation
- Control (Active Comparator): Standard probation - delivered by a standard probation officer - care as usual
  Interventions: Behavioral: Specialty Mental Health Probation

INTERVENTIONS:
Behavioral: Specialty Mental Health Probation — Specialty mental health probation includes the following components: (1) exclusively mentally ill caseload of probationers; (2) reduced caseload of 40-45 probationers; (3) problem-solving supervision orientation; (4) ongoing training and consultation; and (5) greater connection with local mental health services

SUMMARY:
Specialty mental health probation for offenders with severe mental illness has been widely disseminated; however, randomized studies are needed to determine its effectiveness. The purpose of the study is to test the feasibility and efficacy of specialty mental health probation (SMHP) for probationers with mental illness in North Carolina. 320 adult probationers with mental illness in will be randomly assigned to specialty mental health probation (experimental condition) or usual probation (control condition). Probationers assigned to the experimental condition will be supervised by specialty mental health probation officers, who will have reduced caseloads and advanced training in mental health and other topics. Probationers assigned to the control condition will receive standard probation. Criminal justice and mental health outcomes will be examined.

DETAILED DESCRIPTION:
Specialty mental health probation for offenders with severe mental illness has been widely disseminated; however, randomized studies are needed to determine its effectiveness. The purpose of the study is to test the feasibility and efficacy of specialty mental health probation (SMHP) for probationers with mental illness in North Carolina. 320 adult probationers with severe mental illness in will be randomly assigned to receive specialty mental health probation (experimental condition) or standard probation (control condition). Probationers assigned to the experimental condition will be supervised by specialty mental health probation officers, who will have reduced caseloads and advanced training in mental health and other topics. Probationers assigned to the control condition will receive standard probation. Criminal justice and mental health outcomes will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Qualifying diagnosis of severe mental illness - schizophrenia, bipolar disorder, major depression, post-traumatic stress disorder + on probation in North Carolina + capable of passing study competency quiz administered by the research team

Exclusion Criteria:

* None

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 311 (Actual)
Dates: Start 2016-09-22 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Recidivism | 24 months
  Recidivism, probation revocation or other criminal justice events

SECONDARY OUTCOMES:
Mental health service engagement | 24 months
  Administrative data from local and state mental health authorities will be accessed to assess mental health service utilization
Mental health functioning | 6 months
  Assessment of mental health functioning - standardized measure (Symptom Checklist - SCL-10-R)
Social support | 6 months
  Assessment of social support - standardized measure (Medical Outcomes Study - Social Support Scale [MOS])
Life events checklist | Baseline
  Assessment of traumatic life events - standardized measure (Life Events Checklist - LEC-5 Standard)
Substance use | 24 months
  Criminal justice contact related to substance use - via administrative records
Social network (researcher-created measure of social support network) | 6 months
  Access and utilization of pro-social network as measured by a researcher-created instrument
Dual Role Relationship Inventory (DRRI, standardized measure) | baseline, 6 months
  Assessment of probationer's relationship with probation officer

CONTACTS AND LOCATIONS:
Overall Officials: Gary Cuddeback, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No